CLINICAL TRIAL: NCT06992206
Title: What Lies Beneath the Stone? Metabolic Insights From Composition-based Analysis of Kidney Stones
Acronym: Kidney stone
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Prof.Dr, Hisar Intercontinental Hospital
Other Study IDs: Hisar-KSD-2025-33
Record Dates: First submitted 2025-05-18; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Urolithiasis, Calcium Oxalate
Keywords: Calcium oxalate; Metabolic evaluation; Urolithiasis; Stone composition
MeSH Terms: conditions — Nephrolithiasis, Calcium Oxalate; Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First-time Stone Formers: Adult patients who presented with their first episode of kidney stone disease. These patients underwent stone composition analysis via FTIR spectroscopy and metabolic evaluation including serum and 24-hour urine testing to identify risk factors for initial stone formation.
  Interventions: Other: Metabolik taş analizi ile retrospektif gözlem
- Recurrent Stone Formers: Patients with a documented history of recurrent kidney stone episodes. These individuals were evaluated to assess differences in metabolic profiles and stone composition compared to first-time stone formers, with the aim of identifying predictors of recurrence and optimizing preventive strategies.
  Interventions: Other: Metabolik taş analizi ile retrospektif gözlem

INTERVENTIONS:
Other: Metabolik taş analizi ile retrospektif gözlem — This study did not involve an active intervention. It retrospectively analyzed medical records of 506 patients who underwent compositional analysis of kidney stones to identify metabolic abnormalities. The aim was to evaluate stone composition in relation to metabolic parameters such as serum and 24-hour urine values, without modifying patient treatment.
  Other Names: Böbrek taşı kompozisyonu değerlendirmesi Retrospektif metabolik değerlendirme

SUMMARY:
This retrospective observational study investigates the metabolic abnormalities associated with different types of kidney stones by analyzing their composition. The study includes adult patients diagnosed with urolithiasis, whose stone samples were analyzed using Fourier Transform Infrared (FTIR) spectroscopy. Clinical, biochemical, and 24-hour urine metabolic parameters were compared between first-time and recurrent stone formers, and among subtypes of calcium oxalate stones (monohydrate vs. dihydrate). The goal is to identify metabolic risk factors that contribute to stone formation and recurrence, and to provide insights for individualized prevention strategies.

DETAILED DESCRIPTION:
This retrospective study aims to evaluate the metabolic characteristics of patients with urolithiasis based on kidney stone composition. Data were collected from patients treated for kidney stones between January 2010 and December 2024 at a tertiary urology center. Stone analysis was performed using FTIR spectroscopy, classifying stones into subtypes including calcium oxalate monohydrate (COM), calcium oxalate dihydrate (COD), uric acid, and mixed types.

Serum levels of calcium, phosphorus, uric acid, creatinine, and parathyroid hormone (PTH), along with 24-hour urine values (calcium, oxalate, citrate, uric acid, volume, and pH), were recorded. The study primarily compares metabolic differences between:

First-time vs. recurrent stone formers

COM vs. COD stone subtypes

Findings from this study are expected to improve understanding of metabolic risk factors and contribute to the development of tailored metabolic evaluations and dietary or pharmacological preventive strategies for recurrent stone formers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients diagnosed with kidney stones between January 2010 and December 2024
* Stone composition analyzed via Fourier-transform infrared (FTIR) spectroscopy
* Available metabolic panel including serum and 24-hour urine values

Exclusion Criteria:

* Patients with secondary hyperparathyroidism, renal tubular acidosis, or other systemic metabolic diseases affecting stone formation
* Patients with incomplete medical records
* Patients with non-calcium-based stones (e.g., uric acid, struvite, cystine)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study included 506 patients who presented with nephrolithiasis and underwent metabolic evaluation of stone composition. Data were collected retrospectively from medical records at Hisar Intercontinental Hospital between 2010 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Kalsiyum oksalat taşı tipine göre serum ve 24 saatlik idrar parametrelerinin dağılımı Zaman Çerçevesi (Time Frame): 01 Ocak 2010 - 31 Aralık 2024 tarihleri arasında toplanan hasta verileri | January 2010 and December 2024
  FTIR spektroskopisi ile taş bileşimi belirlenen hastalar arasında, kalsiyum oksalat monohidrat (COM) ve dihidrat (COD) taşı olan bireylerin metabolik parametreleri (serum kalsiyum, fosfor, magnezyum, parathormon; 24 saatlik idrarla kalsiyum, oksalat, sitrat, pH, Na, ürik asit vb.) retrospektif olarak analiz edilmiştir.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared include stone composition types (e.g., calcium oxalate monohydrate vs dihydrate), serum metabolic parameters (e.g., calcium, phosphorus, PTH), and 24-hour urine findings (e.g., oxalate, citrate, pH, sodium, uric acid).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available 6 months after publication of the main study results and will remain accessible for a period of 36 months upon request.
Access Criteria: Qualified researchers affiliated with academic or healthcare institutions may request access to the de-identified IPD for secondary analysis or meta-analysis. Requests should be submitted to the corresponding author with a detailed research proposal. Data access will be granted following review and under a data-sharing agreement.